CLINICAL TRIAL: NCT05710926
Title: A Confirmatory Randomized Controlled Trial Comparing Evolutionary Systems Therapy for Schizotypal Personality Disorder With Cognitive Behavioral Therapy
Brief Title: Evolutionary Systems Therapy for Schizotypy
Acronym: ESTS-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tages Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESTS-23
Record Dates: First submitted 2023-01-17; First posted 2023-02-02 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Schizotypal Personality Disorder
Keywords: compassion; metacognition; personality disorder; schizotypy
MeSH Terms: conditions — Schizotypal Personality Disorder; Personality Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants are randomly assignedon a 1:1 ratio to one of two groups in parallel for the duration of the study. Each participant will access a talk therapy lasting 6 months (24 weekly sessions).
Who Masked: Investigator, Outcomes Assessor
Masking Description: An experienced first clinician will make the initial assessment without knowing the assignment to the two groups. Similarly, a second expert clinician will evaluate the participants at the end of th.e intervention without knowing the assignment to the two groups. The data will then be anonymized and a statistician will analyze them without knowing which group corresponds to which treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Active Comparator): Cognitive Behavioral Therapy for Personality Disorder as manualized by Beck, Davis, Freeman and Beck in their book (2016) will be delivered to partecipants in the active control group.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Evolutionary Systems Therapy for Schizotypy (Experimental): Evolutionary Systems Therapy for Schizotypy as manualized by Cheli and colleagues in their trial (2023) will be delivered to partecipants in the experimental group.
  Interventions: Behavioral: Evolutionary Systems Therapy for Schizotypy

INTERVENTIONS:
Behavioral: Evolutionary Systems Therapy for Schizotypy — A novel therapy for schizotypal traits integrating evolutionary psychopathology, compassion focused therapy, and metacognitively oriented psychotherapy.
  Arms: Evolutionary Systems Therapy for Schizotypy
Behavioral: Cognitive Behavioral Therapy — An adaptation of Cognitive Behavioral Therapy for those diagnosed with personaloty disorders.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
This study aims at replicating existing preliminary evidence about the effectiveness of Evolutionary Systems Therapy for Schizotypy (ESTS). The present randomized controlled trial (RCT) will compare ESTS with Cognitive Behavioral Therapy (CBT) in treating Schizotypal Personality Disorder (SPD). The main questions our RCT aims to answer are:

1. Is ESTS more effective than CBT in treating SPD?
2. Is ESTS more feasible than CBT in treating SPD?

38 patients diagnosed with SPD will be recruited and randomly allocated to either the experimental group (i.e. ESTS) or the control group (CBT). Primary outcome will be reduction in general symptomatology, whereas secondary outcomes will be changes in target mechanisms (self-criticism and metacognition) and remission from diagnosis.

DETAILED DESCRIPTION:
A previous study suggested how ESTS (experimental group; EG) may be not inferior in respect to a combine treatment comprising of CBT and psychopharmacological treatment (control group; CG). Despite the encouraging results, it has been suggested that the presence in the CG of a mandatory pharmacological treatment would have represented a bias. Indeed, a few partecipants refused pharmacological treatment.

Thus, the investigators outlined an RCT aimed at comparing the two interventions (ESTS and CBT) without any mandatory pharmacological treatment. Moreover, the investigators consider the need for a pharmacological treatment during the study as an exclusion criterion.

The investigators expect to extend our knowledge about the feasbility and effectiveness of ESTS for those diagnosed with SPD:

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizotypal Personality Disorder at SCID-5-AMPD Module III
* Age 18 or older
* Being capable of reading and signing the inform consent form in Italian
* Being capable of attending a talk therapy in Italian

Exclusion Criteria:

* Being diagnosed with schizophrenia spectrum disorders or other psychosis disorder
* Being diagnosed with neurodevelopmental or neurological disorders
* Being diagnosed with bipolar disorder
* Being under any psychological or pharmacological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in general symptomatology | 2 measurements: one at baseline assessment; one at final assessment
  Change in the total score of Symptom Checklist-90-R (SCL-90-R) between two measurements

SECONDARY OUTCOMES:
Change in metacognition | 2 measurements: one at baseline assessment (once the intervention starts); one at final assessment (6 months after, that is after weekly scheduled 24 sessions)
  Change in total score of Metacognition Assessment Scale - Abbreviated (MAS-A) between two measurements
Change in critical beliefs about self | 2 measurements: one at baseline assessment (once the intervention starts); one at final assessment (6 months after, that is after weekly scheduled 24 sessions)
  Change in the Hated-self scale of The Forms of Self-Criticizing/attacking and Self-reassuring Scale (FSCRS) between two measurements
Change in critical beliefs about others | 2 measurements: one at baseline assessment (once the intervention starts); one at final assessment (6 months after, that is after weekly scheduled 24 sessions)
  Change in Socially prescribed perfectionism scale of Multidimensional Perfectionism Scale (MPS) between two measurements
Change in schizotypal traits 1 | 2 measurements: one at baseline assessment (once the intervention starts); one at final assessment (6 months after, that is after weekly scheduled 24 sessions)
  Change in Psychoticism scale of Personality Inventory for DSM-5 (PID-5) between two measurements
Change in schizotypal traits 2 | 2 measurements: one at baseline assessment (once the intervention starts); one at final assessment (6 months after, that is after weekly scheduled 24 sessions)
  Change in Detachment scale of Personality Inventory for DSM-5 (PID-5) between two measurements
Change in remission from primary diagnosis | 2 measurements: one at baseline assessment (once the intervention starts); one at final assessment (6 months after, that is after weekly scheduled 24 sessions)
  Change in Diagnosis of Schizotypal Personality Disorders trough Structured Clinical Interview for the DSM-5 Alternative Model for Personality Disorders (SCID-5-AMPD) Module III between two measurements

CONTACTS AND LOCATIONS:
Overall Officials: Simone Cheli, PhD, Principal Investigator — Tages Onlus
Locations (1):
- Centro di Psicologia e Psicoterapia Tages Onlus - Firenze, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data will be anonymized and shared through Open Science Foundation at the end of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol, SAP, and ICF will be shared before the end of February 2023.